CLINICAL TRIAL: NCT07326319
Title: The Effect of Periodontal Treatment on Tongue Coating and Olfactory Functions in Patients With Periodontitis
Brief Title: Effect of Periodontal Treatment on Tongue Coating and Smell Function
Acronym: EPTOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, Gulucag Giray Tekin, Assistant professor, Batman University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BatmanU-PERİO-01-2025
Record Dates: First submitted 2025-12-03; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis; Tongue Coating; Olfactory Dysfunction
Keywords: Periodontitis; Periodontal Treatment; Tongue Coating
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: This is a single-arm, pre-post interventional study designed to evaluate the effects of non-surgical periodontal treatment on tongue coating and olfactory function in patients with periodontitis. All participants receive the same standardized periodontal therapy, and assessments are conducted before treatment (baseline) and three days after the final treatment session. Clinical periodontal parameters (Plaque Index, Gingival Bleeding Index, Probing Pocket Depth, Clinical Attachment Loss), tongue coating (Winkel Tongue Coating Index), and olfactory function (Sniffin' Sticks TDI score) are measured at both time points.
  No randomization or blinding is applied, as all participants receive the same intervention, and each patient serves as their own control.
Masking Description: No parties are masked in this study; it is an open-label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Periodontal Treatment Group (Experimental): Participants in this group receive standard non-surgical periodontal treatment, including scaling and root planing. Clinical periodontal parameters (Plaque Index, Gingival Bleeding Index, Probing Pocket Depth, Clinical Attachment Loss), tongue coating (Winkel Tongue Coating Index), and olfactory function (Sniffin' Sticks TDI score) are measured before treatment (baseline) and three days after the final treatment session. Each participant serves as their own control for pre- and post-treatment comparisons.
  Interventions: Procedure: Non-Surgical Periodontal Treatment (Scaling and Root Planing

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Treatment (Scaling and Root Planing — Participants receive standard non-surgical periodontal treatment, including scaling and root planing of all teeth except third molars. Clinical periodontal parameters-including Plaque Index, Gingival Bleeding Index, Probing Pocket Depth, and Clinical Attachment Loss-are recorded before treatment and three days after the final session. Tongue coating is assessed using the Winkel Tongue Coating Index, and olfactory function is evaluated using the Sniffin' Sticks TDI score. Each participant serves as their own control for pre- and post-treatment comparisons.

SUMMARY:
This study aims to investigate the effect of periodontal treatment on olfactory function in patients with periodontitis by comparing pre- and post-treatment periodontal indices, Winkel tongue coating scores, and Sniffin' Sticks TDI components.

DETAILED DESCRIPTION:
Periodontitis is a multifactorial chronic inflammatory disease caused by dental plaque, characterized by connective tissue destruction, periodontal pocket formation, and alveolar bone loss. Pathogenic bacteria associated with periodontitis and the host inflammatory response contribute not only to periodontal tissue breakdown but also to oral malodor (halitosis) and disruption of the oral microbiota. Progressive periodontal inflammation promotes the formation of a dense biofilm on the dorsum of the tongue, containing bacterial products, keratinized epithelium, and protein residues. This leads to increased tongue coating, which serves as a primary source of volatile sulfur compounds (VSCs) strongly associated with halitosis.

The Winkel Tongue Coating Index (WTCI) is commonly used to assess tongue coating and is an important clinical indicator for both halitosis and periodontal status. The bacterial load on the tongue also acts as a reservoir, contributing to dysbiosis of the oral microbiota in periodontitis patients.

Recent studies have also highlighted a potential relationship between periodontitis and olfactory function. Proinflammatory cytokines released during periodontal inflammation, such as IL-1β, TNF-α, and IL-6, may negatively affect the olfactory epithelium, leading to impaired odor threshold, discrimination, and identification abilities. Olfactory function is commonly evaluated using the Sniffin' Sticks test, which includes three subtests: odor threshold, odor discrimination, and odor identification. The sum of these tests, known as the TDI score, reflects overall olfactory capacity.

Previous studies have shown that periodontal treatment can improve tongue coating and halitosis. However, studies simultaneously evaluating pre- and post-treatment tongue coating indices, periodontal indices, and olfactory function (TDI scores) are limited. The aim of this study is to compare these parameters before and after periodontal treatment in patients with periodontitis and to investigate the effect of periodontal therapy on olfactory function.

This study was approved by the Batman University Interventional Clinical Research Ethics Committee (Approval No: 2024/08-04). All procedures and data collection were conducted in accordance with the Declaration of Helsinki, and all participants provided written informed consent.

Participant Selection and Exclusion Criteria

A total of 108 non-smoking volunteers with periodontitis were included. Inclusion required the presence of at least two teeth with probing pocket depth (PPD) ≥ 5 mm and alveolar bone loss visible on full-mouth radiographs. Exclusion criteria were: current smokers, participants who received periodontal treatment in the last 6 months, pregnant or breastfeeding women, individuals who had received antibiotics in the last 3 months, or those with systemic conditions potentially affecting olfactory function.

Radiographic Periodontal Assessment

Full-mouth orthopantomographic radiographs were obtained to confirm the periodontal diagnosis and assess alveolar bone status for all participants.

Olfactory Function Assessment

Before periodontal treatment (Phase 1), olfactory function was objectively evaluated in all 108 participants using the Sniffin' Sticks test (Burghart Messtechnik, Holm, Germany). This psychophysical test assesses odor threshold, odor discrimination, and odor identification, each scored on a scale from 0 to 16. The sum of these subtests provided the TDI score, reflecting overall olfactory capacity. A second assessment was performed 3 days after the final periodontal treatment session.

Periodontal Measurements

Clinical periodontal parameters-including Plaque Index (PI), Gingival Bleeding Index (GBI), Probing Pocket Depth (PPD), and Clinical Attachment Loss (CAL)-were recorded for all teeth except third molars using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA). Four sites per tooth (mesial, distal, buccal, lingual) were measured. All measurements were performed by a calibrated periodontist (GGT), and post-treatment measurements were repeated 3 days after the final session. Intra-examiner reliability was assessed using the weighted Kappa test, yielding satisfactory values (e.g., 0.82 for PPD).

Tongue Coating Assessment

Digital photographs of the tongue dorsum were taken at a standardized distance of 60 cm, ensuring patient privacy. Images were analyzed at 1680 × 1050 pixels resolution using Adobe Photoshop. The Winkel Tongue Coating Index (WTCI) was applied, dividing the dorsum into six areas (three anterior, three posterior). Each region was scored as: 0.5 - no coating, 1.5 - mild coating, 2.5 - severe coating. Scores from all six areas were summed (range 0-12) to obtain the final tongue coating score. Two calibrated observers (GGT, VE) independently scored all images, and the average was used as the final score for each participant. Inter-rater reliability and reproducibility were confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with a clinical diagnosis of periodontitis
2. At least two teeth with probing pocket depth (PPD) ≥ 5 mm
3. Alveolar bone loss visible on full-mouth radiographs
4. Non-smokers
5. Ability to provide written informed consent

Exclusion Criteria:

1. Current smokers
2. Periodontal treatment within the past 6 months
3. Pregnancy or breastfeeding
4. Antibiotic use within the past 3 months
5. Systemic diseases or conditions known to affect olfactory function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Olfactory Function (TDI Score) Following Periodontal Treatmen | Time Frame: Baseline (before periodontal treatment) and 3 days after the final treatment session
  The primary outcome of this study is the change in olfactory function following non-surgical periodontal treatment. Olfactory function is assessed using the Sniffin' Sticks Test Battery, which consists of three subtests: odor threshold, odor discrimination, and odor identification. The sum of these three subtests yields the TDI score, with a total score ranging from 1 to 48. Higher TDI scores indicate better olfactory function.
  Measurements are performed at baseline, prior to periodontal treatment, and three days after completion of the final treatment session in order to evaluate short-term changes in olfactory function attributable to periodontal therapy. This pre-post comparison allows each participant to serve as their own control.

SECONDARY OUTCOMES:
Change in Tongue Coating Index Score | Baseline (pre-treatment) and 8 weeks after completion of periodontal treatment
  This study evaluates the effects of non-surgical periodontal treatment on tongue coating and olfactory function in patients with periodontitis. A total of 108 non-smoking adults with periodontitis were included. Individuals with recent periodontal treatment, pregnancy or breastfeeding, recent antibiotic use, or systemic conditions affecting olfactory function were excluded.
  All participants received scaling and root planing. Periodontal parameters were recorded at baseline and three days after treatment. Tongue coating was assessed using the Winkel Tongue Coating Index, and olfactory function was evaluated using the Sniffin' Sticks Test Battery (TDI score). Pre- and post-treatment measurements were compared, with each participant serving as their own control.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - batman University Faculty of Dentistry, Department of Periodontology, Batman, Batman City
  - batman University Faculty of Dentistry,, Batman, Batman City

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared due to ethical and privacy considerations, including protection of participant confidentiality and informed consent restrictions.